CLINICAL TRIAL: NCT05990153
Title: Evaluation of the Efficacy of Manual Therapy, Therapeutic Exercise and the Two Modalities Combined in Pain Reduction in Patients Suffering From Cervicogenic Headache, or Primary Headache (Tension-type Headache, Migraine, Trigeminal Autonomic Headache)
Brief Title: Evaluation of the Efficacy of Manual Therapy, Therapeutic Exercise and the Two Modalities Combined in Pain Reduction in Patients With Headache
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Silvia Sterzi, Director of Physical Medicine and Rehabilitative Unit, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023.028
Record Dates: First submitted 2023-05-29; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Headache
Keywords: headache; rehabilitation; manual therapy; exercise
MeSH Terms: conditions — Headache; Motor Activity | interventions — Myofascial Release Therapy; Musculoskeletal Manipulations; Exercise Therapy

STUDY DESIGN:
Intervention Model Description: The allocation sequence will occur by 1:1:1:1 randomization, using the Clinical Trial Randomization tool (web https://ctrandomization.cancer.gov/), stratifying by headache type. The allocation of patients will be hidden, through the use of sealed envelopes in which the randomization will be contained. The enrollment will be carried out by the medical doctors of the Headache and Neurosonology Center clinics of the Campus Bio-Medico University Hospital Foundation, who will communicate the patient's name to a third person external to the study who will assign the patient according to the randomization plan developed.
Who Masked: Outcomes Assessor
Masking Description: the assessor is unaware of the type of treatment the patients have received
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Myofascial Release (MR) + Therapeutic exercise (TE) (Experimental): Patients in the MR+TE group will undergo 12 sessions (3 d/week) of sub-occipital inhibition treatment as a combined muscle and soft tissue inhibition technique. The physiotherapist will apply deep pressure which will be maintained for a total of 10 minutes until the sub-occipital tissues are released. In addition to this technique, the method of pumping and manual treatment (acupressure) of the trigger points on the sub-occipital muscles, on the upper bundles of the trapezius bilaterally, on the sternocleidomastoid bilaterally and on the scalene muscles bilaterally will be applied for a further 10 minutes for a total treatment with myofascial release equal to 20 minutes. At the end of the MR session, the 20-minute TE session will be performed in the same way as described in the TE intervention group.
  Interventions: Other: Myofascial Release (MR); Other: Therapeutic exercise (TE)
- Manual therapy (MT) + Therapeutic exercise (TE) (Experimental): The MT+TE intervention group will carry out rehabilitation treatment with a structured protocol based on mobilizations according to the Mulligan method. Treatment according to Mulligan will be carried out at the discretion of the therapist on the basis of daily evaluations of cervical dysfunction and the eventual manifestation of headache. 5 different techniques will be performed on the patient in 12 sessions (3 v/week, for 4 weeks) as described in Satpute, K., Bedekar, N. & Hall, T. Effectiveness of Mulligan manual therapy over exercise on headache frequency, intensity and disability for patients with migraine, tension-type headache and cervicogenic headache - a protocol of a pragmatic randomized controlled trial. BMC Musculoskelet Disord 22, (2021)..
  Interventions: Other: Manual therapy (MT); Other: Therapeutic exercise (TE)
- Therapeutic exercise (TE) (Experimental): Patients in the TE intervention group will be asked to perform 12 sessions (3 day/week) of TE supervised by a physiotherapist. Each session will have a total duration of 40 min divided into 20 min of aerobic exercise and 20 min of TE. Aerobic exercise consists of a total of 20 min of activity on a stationary bike using parameters to increase performance (intensity over 20 min) progressively based on fatigue (Borg scale).The TE consists of warm-up and cool-down exercises for the cervical ROM, associated with stretching exercises of the cervical and scapulothoracic muscles. After the warm-up, muscle strengthening exercises will be performed (isometric, concentric and eccentric contractions of the cervical muscles).
  Interventions: Other: Therapeutic exercise (TE)
- Control (Active Comparator): Patients assigned to the control group will follow the pharmacological treatment according to medical doctor indications (clinical practice).
  Interventions: Drug: clinical practice drug treatment

INTERVENTIONS:
Other: Myofascial Release (MR) — Myofascial release therapy is a type of gentle, constant massage that releases tightness and pain throughout myofascial tissues.
  Arms: Myofascial Release (MR) + Therapeutic exercise (TE)
Drug: clinical practice drug treatment — drug treatment according to the medical indications of clinical practice
  Arms: Control
Other: Manual therapy (MT) — The manual therapy consists of the concurrent application of sustained accessory mobilization applied by a therapist and an active physiological movement to end range applied by the patient. Passive end-of-range overpressure, or stretching, is then delivered without pain as a barrier.
  Other Names: Mulligan Concept
  Arms: Manual therapy (MT) + Therapeutic exercise (TE)
Other: Therapeutic exercise (TE) — The ET consists of an initial phase of aerobic exercise (cyclette), subsequently the intervention foresees exercises for the cervical ROM, stretching exercises of the cervical and scapulothoracic muscles and muscle strengthening exercises (isometric, concentric and eccentrics of the cervical musculature).
  Arms: Manual therapy (MT) + Therapeutic exercise (TE); Myofascial Release (MR) + Therapeutic exercise (TE); Therapeutic exercise (TE)

SUMMARY:
The study aims to evaluate which is the best approach for the non-pharmacological treatment of patients with different types of primary headaches (tension-type headache (TTC), trigeminal autonomic headache (TACs) and migraine) or cervicogenic headache by comparing three methods of intervention to control treatment (drug therapy): therapeutic exercise (TE), myofascial release + TE, and Mulligan's manual therapy + TE. The efficacy will be evaluated in terms of reduction of headache episodes, pain intensity and its duration.

DETAILED DESCRIPTION:
Patients will be evaluated before the start of treatment (T0), at the end of treatment (T1), 3 months after T1 (T2), 6 months after T1 (T3). Results will be stratified by gender, age range, and type of headache diagnosed.

The 3 non-pharmacological treatment groups will carry out 12 treatment sessions, 3 times a week for 4 weeks, with a duration of 45 minutes each. The control group (CTRL) will carry out pharmacological treatment according to clinical practice, the patients of the CTRL group at the end of the last follow-up evaluation (T3 at 6 months) at their request will be randomized into one of the other three intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from primary headache or cervicogenic headache;
* Age > 18 years;
* signature of the informed consent.

Exclusion Criteria:

* upper cervical spine instability;
* cervical arterial insufficiency
* cervical spine fractures
* pregnancies
* rheumatoid arthritis
* severe cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Headache frequency | 4 weeks (end of treatment)
  number of headache attacks in one month
Headache frequency | 3 months after the end of the treatment
  number of headache attacks in one month
Headache frequency | 6 months after the end of the treatment
  number of headache attacks in one month

SECONDARY OUTCOMES:
Headache clinical presentation | 4 weeks (end of treatment)
  the Visual Analogue Scale corresponds to the visual representation of the amplitude of pain felt by the patient at rest and in movement of the headache symptom. The scale consists in a straight horizontal line of100 mm length. The ends are defined as the extreme limits of the pain, and is orientated from the left (no pain) to the right (worst pain)
Headache clinical presentation | 3 months after the end of the treatment
  the Visual Analogue Scale corresponds to the visual representation of the amplitude of pain felt by the patient at rest and in movement of the headache symptom. The scale consists in a straight horizontal line of100 mm length. The ends are defined as the extreme limits of the pain, and is orientated from the left (no pain) to the right (worst pain)
Headache clinical presentation | 6 months after the end of the treatment
  the Visual Analogue Scale corresponds to the visual representation of the amplitude of pain felt by the patient at rest and in movement of the headache symptom. The scale consists in a straight horizontal line of100 mm length. The ends are defined as the extreme limits of the pain, and is orientated from the left (no pain) to the right (worst pain)
Headache related disability | 4 weeks (end of treatment)
  The headache related disability is assessed through the neck disability index
Headache related Disability | 3 months after the end of the treatment
  The headache related disability is assessed through the neck disability index
Headache related Disability | 6 months after the end of the treatment
  The headache related disability is assessed through the neck disability index
Headache related Disability | 4 weeks (end of treatment)
  The headache related disability is assessed through the migraine disability assessment test.
Headache related Disability | 3 months after the end of the treatment;
  The headache related disability is assessed through the migraine disability assessment test.
Headache related Disability | 6 months after the end of the treatment
  The headache related disability is assessed through the migraine disability assessment test.
Perceived Quality of life | 4 weeks (end of treatment)
  The quality of life is assessed through the Migraine-Specific Quality of Life Questionnaire (MSQ)
Perceived Quality of life | 3 months after the end of the treatment
  The quality of life is assessed through the Migraine-Specific Quality of Life Questionnaire (MSQ)
Perceived Quality of life | 6 months after the end of the treatment
  The quality of life is assessed through the Migraine-Specific Quality of Life Questionnaire (MSQ)
Perceived Quality of life | 4 weeks (end of treatment)
  The quality of life is assessed through the Short Form-36 Health Survey
Perceived Quality of life | 3 months after the end of the treatment
  The quality of life is assessed through the Short Form-36 Health Survey
Perceived Quality of life | 6 months after the end of the treatment
  The quality of life is assessed through the Short Form-36 Health Survey
Cervical Range of Motion | 4 weeks (end of treatment)
  Active cervical range of motion recorded through the dynamo vald system
Cervical Range of Motion | 3 months after the end of the treatment
  Active cervical range of motion recorded through the dynamo vald system
Cervical Range of Motion | 6 months after the end of the treatment
  Active cervical range of motion recorded through the dynamo vald system
Cervical muscles Strength | 4 weeks (end of treatment)
  Peak strength of the neck muscles will be measured with the Dynamo portable dynamometer (VALD Performance, Australia)
Cervical muscles Strength | 3 months after the end of the treatment
  Peak strength of the neck muscles will be measured with the Dynamo portable dynamometer (VALD Performance, Australia)
Cervical muscles Strength | 6 months after the end of the treatment
  Peak strength of the neck muscles will be measured with the Dynamo portable dynamometer (VALD Performance, Australia)
Drug intake | 4 weeks (end of treatment)
  Number of drug intake reported in the headache diary
Drug intake | 3 months after the end of the treatment
  Number of drug intake reported in the headache diary
Drug intake | 6 months after the end of the treatment
  Number of drug intake reported in the headache diary

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Sterzi, MD, Principal Investigator — Fondazione Policlinico Universitario Campus Bio-Medico
Locations (1):
- Rehabilitation Department Fondazione Policlinico Universitario Campus Bio-Medico, Roma, RM, Italy